CLINICAL TRIAL: NCT03776461
Title: Clinical Evaluation of the Safety and Performance of Fractional Radiofrequency for the Treatment and Reduction of Facial Wrinkles
Brief Title: Fractional Radiofrequency for the Treatment and Reduction of Facial Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: VI0918
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Rhytides; Wrinkle
Keywords: fractional radiofrequency; fractional RF; facial wrinkles; wrinkles

STUDY DESIGN:
Intervention Model Description: Prospective, single centre, evaluator-blind study
Who Masked: Outcomes Assessor
Masking Description: Evaluator blinded assessment of photographs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 80-pin applicator (Experimental): 3 treatments with the 80-pin tip applicator at 0, 4, and 8 weeks.
  Interventions: Device: Venus Viva
- 160 pin applicator (Active Comparator): 3 treatments with the 160-pin tip applicator at 0, 4, and 8 weeks.
  Interventions: Device: Venus Viva

INTERVENTIONS:
Device: Venus Viva — The Venus Viva™ is a non-invasive medical aesthetic device, intended for use in dermatologic and general surgical procedures, requiring ablation and resurfacing of the skin, using the Viva applicator.

SUMMARY:
Prospective, single centre, evaluator-blind study of the safety and performance of fractional radiofrequency (RF) for the treatment and reduction of facial wrinkles.

DETAILED DESCRIPTION:
The study will evaluate 50 treatment sites in subjects requesting treatment of their facial wrinkles. The study will involve three treatments on both sides of the face with 3-5 week intervals between each treatment. Subjects will be followed at 6 and 12 weeks after their last treatment. Analysis will be performed on all subjects who receive at least one treatment

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male or female subjects over 21 years of age who are seeking treatment and reduction of their facial wrinkles.
2. Able to read, understand and voluntarily provide written Informed Consent.
3. Able and willing to comply with the treatment/follow-up schedule and requirements.
4. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment and for the duration of the study and have a negative Urine Pregnancy test at baseline.

Exclusion Criteria:

1. Implantable defibrillators, cardiac pacemakers, and other metal implants
2. Subjects with any implantable metal device in the treatment area
3. Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body (e.g. cochlear implant).
4. Permanent implant in the treated area, such as metal plates and screws, or an injected chemical substance.
5. Current or history of any kind of cancer, or pre-malignant moles.
6. Severe concurrent conditions, such as cardiac disorders.
7. Pregnancy or intending to become pregnant during the study and nursing.
8. Impaired immune system due to immunosuppressive diseases, such as AIDS and HIV, or use of immunosuppressive medications.
9. History of diseases stimulated by heat, such as recurrent herpes simplex in the treatment area; may be enrolled only after a prophylactic regime has been followed for 2 weeks or longer prior to enrollment , or according to Investigator's discretion .
10. Poorly controlled endocrine disorders, such as diabetes.
11. Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
12. History of skin disorders, such as keloids, abnormal wound healing, as well as very dry and fragile skin.
13. History of bleeding coagulopathies, or use of anticoagulants (excluding daily aspirin).
14. Facial dermabrasion, facial resurfacing, or deep chemical peeling within the last three months, if face is treated.
15. Use of isotretinoin (Accutane®) or other retinoids within six months prior to treatment or as per physician's discretion.
16. Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g. ibuprofen-containing agents) one week before and after each treatment session.
17. Any surgical procedure in the treatment area within the last six months or before complete healing.
18. Treating over tattoo or permanent makeup.
19. Excessively tanned skin from sun, tanning beds or tanning creams within the last two weeks.
20. As per the practitioner's discretion, refrain from treating any condition which might make it unsafe for the patient.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Gronski, Study Director — Venus Concept
Locations (1):
- Scripps Clinic Carmel Valley, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 80-pin Applicator: 3 treatments with either the Venus Viva 80-pin or 160-tip applicator at 0, 4, and 8 weeks.
  Venus Viva: The Venus Viva™ is a non-invasive medical aesthetic device, intended for use in dermatologic and general surgical procedures, requiring ablation and resurfacing of the skin, using the Viva applicator.
Period: Overall Study
Arm/Group | 80-pin Applicator
Started | 25
Completed | 18
Not Completed | 7

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Venus Viva: The Venus Viva™ is a non-invasive medical aesthetic device, intended for use in dermatologic and general surgical procedures, requiring ablation and resurfacing of the skin, using the Viva applicator.
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Fitzpatrick Skin Type [Number; unit: participants] — The Fitzpatrick scale is a numerical classification schema for human skin color. Higher numbers mean darker skin.
  participants
    I | 0
    II | 14
    III | 10
    IV | 0
    V | 0
    VI | 0
    Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Subject Satisfaction
Description: Subjects' assessment of satisfaction with the treatment using a 5 point Subject Satisfaction Scale (0=Very Unsatisfied, 4=Very Satisfied) at 6 weeks and 12 weeks post-treatment.
Time Frame: 12 Weeks Post Last Treatment (Around Week 20)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Subjects: 3 treatments with Viva at 0, 4, and 8 weeks. Assessment at Week 20.
  Venus Viva: The Venus Viva™ is a non-invasive medical aesthetic device, intended for use in dermatologic and general surgical procedures, requiring ablation and resurfacing of the skin, using the Viva applicator.
Arm/Group | All Subjects
Number analyzed (Participants) | 18
score on a scale | 2.8 (0.8)

2. Primary Outcome: Subject Satisfaction
Description: as for outcome 1
Time Frame: 6 Weeks Post Last Treatment (Around Week 14)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Subjects: 3 treatments with Viva at 0, 4, and 8 weeks. Assessment at Week 14.
  Venus Viva: The Venus Viva™ is a non-invasive medical aesthetic device, intended for use in dermatologic and general surgical procedures, requiring ablation and resurfacing of the skin, using the Viva applicator.
Arm/Group | All Subjects
Number analyzed (Participants) | 18
units on a scale | 2.6 (0.8)

3. Secondary Outcome: Subject Scale - Visual Analog Scale for Pain
Description: Subject's assessment of discomfort and pain after treatments as measured by a 10 cm visual analog scale (VAS) with 0 being no pain and 10 being pain as bad as it can be. For each subject, the mean VAS score was taken from the 3 treatments.
Time Frame: Post Treatment at the Baseline, 4 Week and 8 Week treatment visits
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Subjects: 3 treatments with Viva at 0, 4, and 8 weeks. Assessment immediately post-treatment.
  Venus Viva: The Venus Viva™ is a non-invasive medical aesthetic device, intended for use in dermatologic and general surgical procedures, requiring ablation and resurfacing of the skin, using the Viva applicator.
Arm/Group | All Subjects
Number analyzed (Participants) | 25
units on a scale | 3.8 (2.4)

4. Secondary Outcome: Subject Scale - 5 Point Scale for Treatment Tolerability With 0 Being Very Intolerable and 4 Very Tolerable.
Description: Subject's assessment of treatment tolerability as measured by a 5-point scale. For each subject the mean of tolerability results from the 3 treatments was taken.
Time Frame: Post Treatment at the Baseline, 4 Week and 8 Week treatment visits
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- All Subjects: 3 treatments with Viva at 0, 4, and 8 weeks. Assessment immediately post-treatment
  Venus Viva: The Venus Viva™ is a non-invasive medical aesthetic device, intended for use in dermatologic and general surgical procedures, requiring ablation and resurfacing of the skin, using the Viva applicator.
Arm/Group | All Subjects
Number analyzed (Participants) | 25
score on a scale | 3.1 (0.8)

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 5/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 2/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=25)
Cold Sore (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT03776461/Prot_SAP_000.pdf